CLINICAL TRIAL: NCT05380297
Title: Validación Del método de análisis Automatizado Del Habla "AcceXible" Para la detección Temprana y Seguimiento de Pacientes Con Deterioro Cognitivo Leve o Demencia en atención Primaria.
Brief Title: Validation of acceXible's Automated Speech Analysis Method for the Early Detection and Monitoring of Patients With Mild Impairment or Dementia in Primary Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Accexible (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PS2020056
Record Dates: First submitted 2022-03-29; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Speech analysis — Speech analysis to detect and monitor mild cognitive impairment

SUMMARY:
Dementia, especially dementia caused by Alzheimer's disease, is considered one of the most severe health problems of our time. It is currently known that the disease begins many years before clinical symptoms appear. The sooner the patient is diagnosed, the sooner the patient will be in a position to prevent further deterioration.

A recent orientation is the analysis of language in relation to the description of images with a high and varied semantic and emotional content. It can be studied that changes in the description of an image check if these changes are associated with the evolution of a person with probable impairment both in memory and cognitive as well as emotional, psychiatric, behavioral and even in their interaction with environmental factors especially those associated with socialization and loneliness.

Thus, the purpose of this study is to validate speech analysis AI models.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 55+ years of age with suspected MCI or diagnosis of dementia and obtains a score greater than 20 on the MMSE.
* Patients must have agreed to participate in the study and have voluntarily signed the informed consent.
* (Healthy) Participants without a diagnosis neurological, or psychiatric disorders. Or taking medication that can affect cognitive abilities.

Exclusion Criteria

* To have received a diagnosis of a significant psychiatric disorder or other cognitive impairment not due to neurodegeneration.
* To have significant vision problems that would affect the ability to perceive visual stimuli.
* To have significant hearing problems that would affect the ability to understand verbal cues.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Vocal biomarkers to assess pre-post variability of normal, MCI and dementia at both point of the study. | Change from the baseline cognitive function at 9 months.
  Standard deviation of normal subjects, MCI and dementia to measure variations in language by using vocal biomarkers.

SECONDARY OUTCOMES:
Correlation between standard cognitive test (MMSE) and linguistic variables obtained by vocal biomarkers. | Through study completion, an average of 1 year.
  With a 95% confidence interval, the correlation between standard cognitive test (MMSE score) and each of the linguistic variables is quantified.

OTHER OUTCOMES:
Change of economic implications of accexible's use in a primary care center. | Through study completion, an average of 1 year.
  Percentage of expenditure when using the platform.

CONTACTS AND LOCATIONS:
Locations (1):
- País Vasco, País Vasco, Basque Country, Spain

IPD SHARING:
Plan to Share IPD: No